CLINICAL TRIAL: NCT05731440
Title: Fluselenamyl - Beta Amyloid PET Imaging for Alzheimer Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology and Neurological Surgery, Washington University School of Medicine
Other Study IDs: Fluselenamyl (FSA)
Record Dates: First submitted 2023-01-03; First posted 2023-02-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy participants: Drug: [18F]-Fluselenamyl. A dosage range of 10 mCi +/- 20% of Fluselenamyl will be injected by a PET certified medical professional followed by 10 ml 0.9% sodium chloride (normal saline) flush.
  Drug: [11C]-Pittsburgh Compound ([11C]PIB) A dosage range between 6.0-20.0 mCi is planned. A PET certified professional will prepare and administer the [11C]-PIB tracer. Participants will receive the PIB injection followed by 10 ml 0.9% sodium chloride (normal saline) flush.
  Interventions: Drug: 18F-Fluselenamyl
- Participants with mild cognitive impairment: Drug: [18F]-Fluselenamyl. A dosage range of 10 mCi +/- 20% of Fluselenamyl will be injected by a PET certified medical professional followed by 10 ml 0.9% sodium chloride (normal saline) flush.
  Drug: [11C]-Pittsburgh Compound ([11C]PIB) A dosage range between 6.0-20.0 mCi is planned. A PET certified professional will prepare and administer the [11C]-PIB tracer. Participants will receive the PIB injection followed by 10 ml 0.9% sodium chloride (normal saline) flush.
  Interventions: Drug: 18F-Fluselenamyl

INTERVENTIONS:
Drug: 18F-Fluselenamyl — Participants will receive a single intravenous bolus injection of 10 mCi ± 20% of the investigational radiotracer 18F-Fluselenamyl and will undergo an 18F-Fluselenamyl PET/CT scan.

SUMMARY:
The purpose of this research study is to determine the safety of a radiotracer 18F-Fluselenamyl using positron emission tomography (PET) imaging.

The investigators will first complete whole-body PET dosimetry studies in healthy adult normal volunteers to calculate the actual radiation dose of each human organ and determine the allowable dose for a human subject when receiving a single dose for a PET scan.

Second, imaging of the brain and neck will be completed in a wide range of ages of healthy adult normal control participants and participants with mild cognitive impairment, both male and females to characterize 18F-Fluselenamyl uptake in the brain, its binding to beta-amyloid plaques, and radiolabeled metabolite will be completed. Amyloid is a protein related to dementia of Alzheimer's disease. 11C-PIB PET imaging along with MRI will also be completed in the same participants and the data will be compared with 18F-Fluselenmayl. 11C-PIB and 18F-Fluselenamyl both bind to beta-amyloid plaques.

Finally, a comparison of the normal control participants to patients with Alzheimer's disease will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, any race
* Age ≥ 18 years
* Healthy volunteers or volunteers with Alzheimer's disease

Exclusion Criteria:

* Has hypersensitivity to 18F-Fluselenamyl or any of its excipients ;
* Has hypersensitivity to 11C-PIB or any of its excipients ;
* Incapable of providing written informed consent or lacking a legally authorized representative (LAR) to provide informed consent ;
* Unwilling or unable to undergo PET scans tracer injections ;
* Unwilling or unable to undergo MRI (Aim 2 and Aim 3);
* Any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data (e.g., renal or liver failure, advanced cancer);
* Women who are currently pregnant or breast-feeding;
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1: Dosimetry - 8 healthy adult normal volunteers (4 Males, 4 Females) will undergo whole-body PET/CT imaging for assessing the safety, dosimetry, and metabolism of 18F-Fluselenamyl.
  Aim 2: Proof of Concept- 36 participants (18 healthy and 18 participants with mild cognitive decline)will undergo 18F-Fluselenamyl imaging of the brain and neck, 11C-PIB imaging of the brain and neck, MRI, and Cognitive testing.
  Aim 3: Performance group- Aim 2 participants will be invited for additional imaging.
  Aim 3A- 10 participants from Aim 2 will undergo repeat 18F-Fluselenamyl imaging ~ 1 month after baseline imaging Aim 3B- 18 participants from Aim 2 will have a longitudinal follow-up visit ~ 18 months after the initial study. They undergo repeat 18F-Fluselenamyl, 11C-PIB, MRI, and Cognitive testing.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of the tracer [18F]-Fluselenamyl for PET Imaging. | 1 year
  Whole-body PET/CT images (skull vertex to proximal thighs) will be obtained in 8 healthy volunteers (4 males and 4 females) for up to a maximum of 4.5 hours immediately following intravenous (IV) injection of 10 mCi ± 20% of [18F]-Fluselenamyl (dosage range calculated from rodent dosimetry data extrapolated to humans).
  The primary objective is to evaluate the biodistribution, kinetics and calculate human dosimetry of this radioligand and confirm it's lack of toxicity in human subjects.
PET imaging of [18F]-Fluselenamyl in healthy normal control participants and human participants with mild cognitive impairment of Alzheimer's dementia. | 2 years
  To assess the sensitivity of [18F]-Fluselenamyl to image Amyloid beta in the setting of mild cognitive impairment, and conduct comparative analysis of PET imaging data using [11C]-PIB imaging in same participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States